CLINICAL TRIAL: NCT03475849
Title: Effects of Gastric Bypass Surgery on Bile Acid Homeostasis
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Carsten Dirksen, MD, PhD, Hvidovre University Hospital
Other Study IDs: GAL-CAJ-16
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: Roux-en-Y Gastric Bypass Surgery; Bile Acid Circulation; Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- RYGB subjects: Morbidly obese patients who has undergone an uncomplicated gastric bypass surgery more than 12 months before study start.
- Control subjects: Age, sex and BMI-matched healthy controls
- SG subjects: Morbidly obese patients who has undergone an uncomplicated sleeve gastrectomy surgery more than 12 months before study start.

SUMMARY:
The purpose of this study is to determine whether the bile acid circulation is changed after gastric bypass surgery. Further, to account for how the changed anatomy of the gut influences how the bile acid and food is mixed in the gut and how this is associated with the changes in gut hormone release after the surgery.

Our hypothesis is that bile acid reabsorption from the gut is increased as animal models suggest so and bile acid blood concentration increases after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 65 years
* For patients: uncomplicated Roux-en-Y Gastric Bypass surgery more than 12 months before study initiation
* For controls: Age, BMI and gender matched with patient group

Exclusion Criteria:

* Previous removal of gall bladder or other abdominal surgeries except appendectomy (and gastric bypass surgery for patient group)
* Known liver disease or thyroid disease requiring antithyroid medication
* Chronic gastrointestinal symptoms
* Any chronic disease interfering with, or susceptive of interfering with appetite or gastrointestinal function
* Any medication interfering with, or susceptive of interfering with appetite or gastrointestinal function
* Smoking within the last month
* Alcohol consumption above 168 grams per week
* Currently pregnant or breast-feeding
* Anaemia with haemoglobin <6,5 mmol/L (<117 mg/dl)
* Loss or gain of more than 3 kg within the last 3 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited from the population undergoing gastric bypass surgery at Hvidovre Hospital (Denmark) Controls are recruited from www.forsoegsperson.dk (Danish webpage for recruitment of trial persons). Controls are recruited by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Differences in time from food intake to mix of food in the gut with bile acid between patients and controls | Patients: >12 months after Gastric Bypass Surgery
Percentage of orally ingested exogenic bile acid that is retained in the body after 7 days | Patients: >12 months after Gastric Bypass Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology at Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark